CLINICAL TRIAL: NCT04823208
Title: A Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3437943 in Japanese Participants With Type 2 Diabetes Mellitus
Brief Title: A Study of LY3437943 in Japanese Participants With Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 17609; J1I-JE-GZBC (Other: Eli Lilly and Company)
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LY3437943 (Experimental): LY3437943 administered subcutaneously (SC)
  Interventions: Drug: LY3437943
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3437943 — Administered SC
  Arms: LY3437943
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The main purpose of this study is to learn about the side effects of LY3437943 when given to Japanese participants with type 2 diabetes mellitus. Blood tests will be performed to investigate how the body processes the study drug and how the study drug affects the body. Each enrolled participant will receive injections of LY3437943 or placebo given just under the skin. For each participant, the study will last up to 5 months, inclusive of screening and will include 16 visits to the study center.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus (T2DM) diagnosed for at least 1 year.
* Have glycated hemoglobin (HbA1c) value ≥ 7.0% and ≤10.0% for participants treated with diet and exercise or HbA1c ≥ 6.5% and ≤ 9.0% for participants who have washed out antidiabetic medications at lead-in and screening
* Have a body mass index (BMI) within the range 23 to 35 kilograms per square meter (kg/m²), inclusive, and a body weight of at least 54 kilograms (Kg).
* Males and females not of childbearing potential

Exclusion Criteria:

* Have type 1 diabetes mellitus (T1DM)
* Have uncontrolled diabetes defined as an episode of ketoacidosis or hyperosmolar state requiring hospitalization
* Have had an episode of severe hypoglycemia, as defined by the occurrence of neuroglycopenic symptoms requiring the assistance of another person for recovery, or have a history of hypoglycemia unawareness or poor recognition of hypoglycemic symptoms.
* Have a history of acute or chronic pancreatitis or fasting serum triglyceride level of >500 milligram per deciliter (mg/dL).
* Have known liver disease, obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or have elevations in aminotransferases (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]) greater than 3× upper limit of normal (ULN).

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-06-23 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 106
  A summary of SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3437943 | Predose on Day 1 through Day 81
  PK: Cmax of LY3437943
PK: Area Under the Concentration Versus Time Curve (AUC) of LY3437943 | Predose on Day 1 through Day 81
  PK: AUC of LY3437943
Change from Baseline in Mean Daily Plasma Glucose (PG) | Baseline through Day 80
  Change from baseline in mean daily PG from 6-point PG profile
Change from Baseline in Glycated Hemoglobin (HbA1c) | Baseline through Day 78
  Change from Baseline in HbA1c
Change from Baseline in Fasting Glucose | Baseline through Day 78
  Change from Baseline in Fasting Glucose
Change from Baseline in Body Weight | Baseline through Day 78
  Change from Baseline in Body Weight

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- Japan (4):
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - P-one clinic, Hachiōji, Tokyo
  - Clinical Research Hospital Tokyo, Shinjuku-ku, Tokyo
  - Yokohama Minoru Clinic, Yokohama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY3437943 in Japanese Participants With Type 2 Diabetes Mellitus (T2DM) — https://trials.lilly.com/en-US/trial/283676